CLINICAL TRIAL: NCT01065870
Title: Phase II Study: Neoadjuvant Gemcitabine, Docetaxel and Capecitabine Followed by Neoadjuvant Radiation Therapy With Gemcitabine and Capecitabine in the Treatment of Stage II and III Pancreatic Adenocarcinoma
Brief Title: Neoadjuvant GTX With Chemoradiation for Pancreatic Cancer (Stage II/III)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, William Sherman, Associate Professor of Clinical Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAD6491
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Cancer Stage II; Pancreatic Cancer Stage III
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): Patients with only venous involvement Treated with 6 cycles og GTX and then surgery
  Interventions: Drug: Neoadjuvant gemcitabine, capecitabine, and docetaxel
- Group II (Experimental): Patients with arterial involvement and may have venous involvement with tumor treated with 6 cycles of GTX, thenb GX/RT and then surgery
  Interventions: Drug: Gemcitabine, capecitabine, docetaxel followed by radiotherapy

INTERVENTIONS:
Drug: Neoadjuvant gemcitabine, capecitabine, and docetaxel — 6 cycles of gemcitabine, capecitabine, and docetaxel. One cycle consists of a 2-week regimen followed by one week off.
  Days 1-14: Capecitabine at 1500mg/m2/day divided into two doses given orally with breakfast and dinner.
  Days 4 and 11: Gemcitabine at 750mg/m2 over 75 minutes IV followed by docetaxel at 30mg/m2 over 30 minutes IV with 10mg of dexamethasone IV prior to treatment.
  Other Names: Gemzar; Xeloda; Taxotere
  Arms: Group I
Drug: Gemcitabine, capecitabine, docetaxel followed by radiotherapy — 6 cycles of gemcitabine, capecitabine, and docetaxel. One cycle consists of a 2-week regimen followed by one week off.
  Days 1-14: Capecitabine at 1500mg/m2/day divided into two doses given orally with breakfast and dinner.
  Days 4 and 11: Gemcitabine at 750mg/m2 over 75 minutes IV followed by docetaxel at 30mg/m2 over 30 minutes IV with 10mg of dexamethasone IV prior to treatment.
  Radiotherapy should start 2 to 3 weeks after last planned dose of GTX. Gemcitabine at 750mg/M2 days 5, 12, 26, 33 along with capecitabine 1000 mg bid for 5 days darbepoetin 200ug, every 2 weeks if the hemoglobin is less than 10.5 gms/dl while undergoing radiotherapy.
  Pegfiligastrim 6mg at the end of week 2 if the WBC count is less than 2500 cells/cu mm.
  Other Names: Gemzar; Taxotere; Xeloda
  Arms: Group II

SUMMARY:
This study is for patients with locally advanced pancreatic cancer (cancer that involves the local blood vessels so it cannot be removed without cutting major blood vessels) that cannot be treated with surgery. The purpose of this study is to assess the safety and benefit of 6 three week cycles of chemotherapy treatment consisting of gemcitabine, capecitabine and docetaxel (also called 'GTX'). The patients fall into two groups. Group I are those with only venous involvement. Group II patients have arterial involvement and may also have venous involvement. If there is arterial involvement, GTX will be followed by 5 and 1/2 weeks of radiation therapy with gemcitabine and capecitabine. After the chemotherapy and radiation treatment, participants may be able to have surgery to remove any remaining pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas (When possible the tissue should be evaluated for K-ras mutation and the patient evaluated for BRCA and p16 mutations.)
* Locally advanced disease determined by Endoscopic ultrasound, CT scan (chest/abdomen/pelvis with contrast), MRI scan (of abdomen with gadolinium) or PET scan.
* No evidence of metastatic disease by CT scan (chest/abdomen/pelvis with contrast), MRI scan (of abdomen with gadolinium) or PET scan.
* Unresectable tumor. (this reflects those patients whose tumors abut, invade or surround a major vessel, either venous or arterial or both)
* No prior chemotherapy or radiation therapy.
* Ineligible for other high priority national or institutional studies.
* Negative serum or urine β-HCG within 1 week of starting treatment for non-pregnant, non-menopausal females.
* Must not have other underlying medical conditions that would make them ineligible for surgery, radiation therapy, or chemotherapy.
* Complete Blood Count and Complete Metabolic Profile:

Absolute Neutrophil Count > 1,500 μl White Blood Count > 3,000/μl Platelet count > 100,000/μl BUN < 1.5 x normal Creatinine < 1.5 normal Hemoglobin > 8.0 g/dl Serum Albumin > 3 mg/dl Total Bilirubin < 3.0 mg/dl SGOT, SGPT, Alkaline Phosphatase < 2.5 x ULN

* Informed consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the nature of this therapy, alternatives, potential benefits, side-effects, risks, and discomforts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2009-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of neoadjuvant regimen of GTX on the 2-year disease free survival rate | 2 years

SECONDARY OUTCOMES:
To describe the effect of neoadjuvant GTX regimen on resectability for those with arterial involvement and those with venous involvement, separately | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Sherman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Sherman WH, Chu K, Chabot J, Allendorf J, Schrope BA, Hecht E, Jin B, Leung D, Remotti H, Addeo G, Postolov I, Tsai W, Fine RL. Neoadjuvant gemcitabine, docetaxel, and capecitabine followed by gemcitabine and capecitabine/radiation therapy and surgery in locally advanced, unresectable pancreatic adenocarcinoma. Cancer. 2015 Mar 1;121(5):673-80. doi: 10.1002/cncr.29112. Epub 2014 Dec 9. PMID 25492104